CLINICAL TRIAL: NCT03569592
Title: Addressing Overdose Risk Among Recently Incarcerated People Living With HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1704005362
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2018-06

CONDITIONS: Drug Overdose Accidental
Keywords: HIV/AIDS; naloxone; incarceration
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Incarcerated people living with HIV/AIDS will be given a brief training on overdose prevention and be given naloxone at discharge from jail.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Overdose Prevention Intervention (Experimental): The experimental group will receive a brief overdose prevention education intervention and be issues naloxone upon discharge from jail.
  Interventions: Behavioral: Overdose Prevention Intervention

INTERVENTIONS:
Behavioral: Overdose Prevention Intervention — Evaluate an overdose prevention education with incarcerated people living with HIV/AIDS.
  Other Names: Addressing Overdose Risk among Recently Incarcerated People Living with HIV/AIDS

SUMMARY:
The overall objective of this study is to evaluate an educational overdose prevention intervention's effectiveness among incarcerated people living with HIV/AIDS, specifically within the context of other outcomes related to health and experiences after incarceration. Results will be used to develop tailored interventions to reduce overdose deaths among high-risk correctional populations.

The research has the following aims:

* Aim 1: Evaluate a pilot program to provide HIV+ inmates with 1:1 overdose prevention training while incarcerated;
* Aim 2: Identify the criminal justice, health, and HIV-related factors associated with overdose risk; and
* Aim 3: Describe the overdose risk experiences of HIV+ former inmates who use opioids after release.

DETAILED DESCRIPTION:
The goal of this research is to establish best practices to address overdose risk in people exiting incarceration, people living with HIV/AIDS (PLWHA), and both populations simultaneously. This contribution is important because this evidence has applications for correctional facilities and HIV clinical practice throughout the United States. The contributions of the proposed pilot study are: to provide evidence on the effectiveness of a targeted intervention on these two high-risk groups, generate exploratory data on predictors of overdose risk specific to HIV status and recent incarceration, and provide context about overdose risk and responses to witnessed overdoses in the first month after release.

In this study, incarcerated PLWHA in the Philadelphia Department of Prisons will be offered overdose training while incarcerated and naloxone (Narcan) at release. Study participants will be given a pre-test on overdose knowledge and attitudes and receive the overdose prevention intervention. Those who are still incarcerated one month later will receive a post-test on overdose knowledge and attitudes. Approximately one month after study participants are released from jail, they will be given a one-month follow-up survey that assesses: overdose knowledge and attitudes (post-test 2), information on personal or witnessed overdoses since release, health and post-incarceration related information, and characteristics of drug use since release. Approximately 20 study participants will participate in a semi-structured interview 4-6 weeks after their release on their experiences with the overdose prevention intervention.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Age 18 and over
* Speaks English
* plans to live in Philadelphia area after release

Exclusion Criteria:

* More than 10 months remaining on a sentence or release date unknown

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Overdose knowledge | time of training until one month after release from jail
  The scale is adapted from the Opioid Overdose Knowledge Scale (OOKS). OOKS subscales measure overdose risks, signs, actions to take in a witnessed overdose, & naloxone use. It has 4 multiple choice questions, 4 forced-choice questions, and 6 true/false statements. Each correct answer is 1 point and incorrect answers are 0. Subscale ranges are 0-9 for overdose risks, 0-10 for signs, 0-11 for actions to take in a witnessed overdose, and 0-15 for naloxone use. The total score range is summed from subscale scores from 0 to 45, with higher scores indicating greater knowledge. The adapted scale assesses the same domains and consists of 4 multiple choice questions, 1 forced-choice question, and 6 true/false statements. Each correct answer is 1 point and incorrect answers are 0. Subscale ranges are 0-5 for overdose risks, 0-4 for overdose signs, 0-5 for overdose actions, and 0-6 for naloxone use. Scores are summed for a total number of 20 points, with higher scores indicating greater knowled
Overdose attitudes | time of training until one month after release from jail
  The scale is adapted from the Opioid Overdose Attitudes Scale (OOAS). OOAS subscales measure overdose response competence (10 items), concerns (8 items), & readiness (10 items). Likert scale options include "Completely Agree", "Agree", "Unsure", "Disagree", and "Completely Disagree" with a score of 1 to 5 assigned to each item. The total score range on the initial measure is summed from the subscales from 28-140 points (1-50 points on subscale competence, 1-40 points on subscale concerns, and 1-50 points on subscale readiness), with higher scores indicating favorable attitudes. The adapted scale also assesses: overdose response competence (4 questions), concerns (3 questions), and readiness (4 questions). Scoring is identical to the full scale, with possible subscales scores ranging from 1-20 for overdose competence, 1-15 for concerns about responding to an overdose, and 1-20 for readiness to respond to an overdose. Scores are summed for a total score range of 11-55. Higher scores in

SECONDARY OUTCOMES:
Witnessed overdoses | 1 month (release from jail until one month after release)
  Information on any witnessed overdoses since release from jail. The domain of witnessed overdoses is not from an existing scale. It is assessed by asking the following: "Have you seen anyone overdose since you left jail? (To be clear, an overdose means someone is unresponsive or cannot be woken up, collapses, has blue skin color, convulsions, difficulty breathing, loses consciousness, or has a heart attack or dies while using drugs.). Answer options are "yes", "no", and "not sure". Those reporting "yes" are directed to a follow-up question: "How many overdoses have you seen since you left jail?" Answer options range include "1", "2", "3", "4", "5 or more". Additional follow-up questions assess the location, response actions of respondent, response actions of others at the scene, and outcome of the overdose for the victim for the most recently witnessed overdose.
Status of naloxone kit | one month after release from jail
  Whether participant was given naloxone at release from jail and where the naloxone kit is at time of follow-up. The domain of "status of naloxone kit" is not from an existing scale. It is assessed by asking: "When you were released from jail, the pharmacy should have given you naloxone. Were you given naloxone?". Answer options include "Yes, I was given a kit when I was released", "I was not given a kit at release but I got one after I was released", "I did not get a kit when I was released and I've never had one", and "Don't know/not sure". Follow-up questions assess where participants received naloxone from if they received a kit after release and the current location of the kit for any respondents reporting having received a naloxone kit at any point and what happened to kits that are no longer in possession of respondents.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States